**Study Title**: Randomized controlled trial to test the feasibility, acceptability, and preliminary effectiveness of a psychosocial intervention to support Alzheimer's family caregivers in Vietnam.

**NCT#**: NCT03587974

Document Date: April 2, 2018

**Document Type**: Informed Consent Form

## Information sheet for verbal consent

- This project is part of a research study to help us test a program to help family members who are caring for someone with memory loss or dementia
- This study is being conducted by the National Geriatric Hospital together with researchers in the United States.
- This is a voluntary study. You are not obligated to participate. There will be no adverse consequence if you choose not to participate.
- If you agree to participate, you will be assigned to one of two groups. One group
  will receive trainings from a healthcare provider who will meet with you 3-6 times
  in your home or another location that is convenient to you. During our meetings,
  you will receive information and training to help you learn more about your
  relative's condition, about how to provide better care, and how to improve your
  own health and well-being.
- The second group will receive educational materials to help care for someone with memory loss and an educational training at the of the study.
- Participants in both groups will also meet two times to answer questionnaires about their health and the care they provide
- We will also ask you questions about your health and the care you provide to your relative.
- You may experience discomfort or fatigue in answering questions. Some
  questions may be upsetting to respond to. In the intervention, some of the
  discussion topics may be upsetting to you. A trained interventionist (nurse or
  social worker) will be able to help you should this occur. Also, you can stop at
  any point.
- We will keep your participation in this research confidential. Your name will not appear any of the records and only the research staff will have access to the data we are collecting.
- We will reimburse you \$10 at the end of each study visit.

Please contact Huong Nguyen at (84) 962546833 in Vietnam and (011) 803-777-2215 in the US or Dr. Trong Hung (84) 435764003 if you have any questions.